CLINICAL TRIAL: NCT01577602
Title: Standard Medication Reconciliation Protocol in the Primary Care Office-based Setting: A Focused Investigation of Two Interventions
Brief Title: Standard Medication Reconciliation Protocol in the Primary Care Office-based Setting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, John Hickner, Professor, The Cleveland Clinic
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Health Services Research
Other Study IDs: 11-667
Record Dates: First submitted 2012-04-12; First posted 2012-04-16 (Estimated); Last update posted 2013-03-14 (Estimated); Status verified 2013-03

CONDITIONS: Medication Reconciliation Between Patients' Self Report and Electronic Medical Record List
Keywords: Medication reconciliation; Self report; Electronic medical record medication list

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Standard practice (No Intervention)
- Printed list intervention (Experimental): Providing patients a list of their current medications before they see medical assistant and begin their visit.
  Interventions: Other: Printed medication list
- Open ended question intervention (Experimental): Medical assistants begin the medication review with a scripted, open ended question (i.e., "tell me about your medications")
  Interventions: Other: Open ended question
- Combined intervention (Experimental)
  Interventions: Other: Combined intervention

INTERVENTIONS:
Other: Printed medication list — Provide a list of patient's current medication list as noted in the EMR
  Arms: Printed list intervention
Other: Open ended question — medical assistants begin medication reconciliation with a scripted open ended question.
  Arms: Open ended question intervention
Other: Combined intervention — Combines the printed medication list with the open ended question
  Arms: Combined intervention

SUMMARY:
The purpose of this study is to determine if two basic medical office visit interventions improve the agreement of medication lists between electronic medical record and patient self, home-based report. The interventions are:

* giving patients a printed list of medications before the visit
* asking the patients about their medications with a scripted, open ended question.

DETAILED DESCRIPTION:
This is a randomized clinical trial of the implementation and initial effectiveness of two interventions for improving medication reconciliation in primary care offices. The interventions we will test are 1) patients reviewing a printed paper copy of their EMR medication list just prior to seeing the physician and 2) medical assistants beginning the interview with an open-ended question. We will test the following two hypotheses:

1. Providing patients a paper copy of their EMR medication list upon check-in, to review for accuracy prior to their office visit, will improve the agreement between the EMR medication list and patient report during a phone interview within one week of the office visit.
2. The medical assistant practice of routinely using an open-ended question to introduce the medication review will improve the agreement between the EMR medication list and patient report during a phone interview within one week of the office visit.

The main outcome measure for this study is full agreement of prescription medications between the medication list in the electronic medical record at the conclusion of patient's office visit and the list generated by pharmacists during a phone interview performed within a week of the office visit.

The study will take place at 2-4 Cleveland Clinic Health Centers in primary care offices. A sample size of 400 patients will be enrolled: 20 pairs of physicians and medical assistants will be invited to volunteer for the study, and 20 patients per MD/MA pair will be recruited. Medical assistants will be trained in using scripted open-ended questions to begin reviewing medications with patients. The study coordinator will implement the printed list intervention by providing a paper list to patients.

Consenting patients will be randomized to one of four groups (A-D):

A: NO patient review of printed medication list & NO open-ended question B: Patient review of printed medication list ONLY C: Open-ended question ONLY D: BOTH patient review of printed medication list & open-ended question

To document the medications that patients report taking, a pharmacist will conduct a detailed phone interview with the patient and/or caretaker within a week of the office visit using a prepared script. The pharmacist will note any discrepancies between the EMR and the patient's/caretaker's self report. In order to be considered in full agreement, the medication list and patient report must agree on the five following elements: 1) name, 2) dose, 3) frequency, 4) route, and 5) PRN status.

Our goal is to statistically test whether the proportion of medication lists in agreement with patient report differs in the intervention group compared to the non-intervention group. First, an unadjusted analysis utilizing a difference of proportions test and linear contrasts as described in the above planned comparisons. Then, a multivariable mixed model will be used to determine the significance of the intervention with adjustment.

If the interventions are successful, they will be incorporated into a standard medication reconciliation protocol for Cleveland Clinic primary care office practice. If highly successful, this protocol could serve as a new standard for medication reconciliation in outpatient primary care practice in the United States.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age
* English speaking
* Current medication list has at least 2 medications listed

Exclusion Criteria:

* less than 18 years of age
* English is not primary language
* Less than 2 medications on medication list

Enrollment only applies to one visit. Patients cannot be enrolled more than one time on the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 424 (Actual)
Dates: Start 2011-10; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Assessment of EMR medication lists and patient report agreement | Within one week of enrolled patient's visit
  To document medications patients report taking, a pharmacist will conduct a detailed phone interview with the patient within a week of the office visit using a prepared script. The pharmacist will note any discrepancies between the EMR and the patient's self report. In order to be considered in full agreement, the medication list and patient report must agree on the five following elements: 1) name, 2) dose, 3) frequency, 4) route, and 5) PRN status.

SECONDARY OUTCOMES:
Assessment of number of medication list discrepancies | Within one week of patients' visit
  Data will be collected in same manner as primary outcome. The secondary outcome focuses on the actual number of discrepancies and what may have caused the discrepancy.

CONTACTS AND LOCATIONS:
Overall Officials: John Hickner, MD, MSc, Study Director — The Cleveland Clinic
Locations (1):
- Cleveland Clinic Foundation, Cleveland, Ohio, United States